CLINICAL TRIAL: NCT05445167
Title: A Phase III Confirmatory Study of KLH-2109 in Uterine Fibroids Patient With Menorrhagia and Pain
Brief Title: A Clinical Study of KLH-2109 in Uterine Fibroids Patient With Menorrhagia and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KLH2302
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-03

CONDITIONS: Uterine Fibroids (MeSH Heading: Leiomyoma)
MeSH Terms: conditions — Leiomyoma | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KLH-2109 (Experimental)
  Interventions: Drug: KLH-2109
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KLH-2109 — Oral administration
  Arms: KLH-2109
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
Multi-center, randomized, double-blind, parallel-group study to confirm superiority of KLH-2109 to placebo in uterine fibroids patient with menorrhagia and pain

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Japanese woman diagnosed with uterine fibroids
* Patients confirmed by transvaginal ultrasonography to have at least 1 myoma that meet all of the following conditions:
* Larger than a certain standard
* No calcification
* Not receiving surgical treatment
* Patients with a normal menstrual cycle
* Patients diagnosed with menorrhagia
* Patients with pain symptoms associated with uterine fibroids

Exclusion Criteria:

* Patients with complication or history of blood system diseases (salasemia, sickle erythrocyte anemia, folic acid deficiency, coagulation disorder, etc.) (excluding iron deficiency anemia and latent iron deficiency anemia)
* Patients with lower abdominal pain due to irritable bowel syndrome or lower abdominal pain due to severe interstitial cystitis
* Patients with undiagnosed abnormal genital bleeding

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a total PBAC score of less than 10 from Week 6 to 12 after beginning of study drug administration | Up to 12 weeks
  PBAC (pictorial blood loss assessment chart) score
Proportion of women with a maximum NRS for pain score of 1 or less during 28 days before the end of study drug administration | Up to 12 weeks
  NRS (numeric rating scale) for pain

SECONDARY OUTCOMES:
Proportion of subjects with a total PBAC score of less than 10 from Week 2 to 6 after beginning of study drug administration | Up to 12 weeks
  PBAC (pictorial blood loss assessment chart) score
Proportion of subjects with a total PBAC score of less than 10 during 6 weeks before end of study drug administration | Up to 12 weeks
  PBAC (pictorial blood loss assessment chart) score
Proportion of subjects with a maximum NRS score of 1 or less for pain symptoms every 28 days | Up to 12 weeks
  NRS (numerical rating scale)
Proportion of subjects with maximum NRS score of zero for pain symptoms during 28 days before end of study drug administration | Up to 12 weeks
  NRS (numerical rating scale)
Proportion of subjects with a maximum NRS score of zero for pain symptoms every 28 days | Up to 12 weeks
  NRS (numerical rating scale)
Average NRS score every 28 days for pain symptoms | Up to 12 weeks
  NRS (numerical rating scale)
Percentage of asymptomatic days (number of the days with NRS score of zero for pain symptoms) during 28 days before end of study drug administration | Up to 12 weeks
  NRS (numerical rating scale)
Percentage of asymptomatic days (number of the days with NRS score of zero for pain symptoms) every 28 days | Up to 12 weeks
  NRS (numerical rating scale)
Incidence of adverse events and adverse drug reactions | Up to 12 weeks
  Adverse events and adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Shimizu, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Clinical Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT05445167/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT05445167/SAP_001.pdf